CLINICAL TRIAL: NCT02006277
Title: A Phase 1, Open-label, Crossover Taste And Pharmacokinetic Study In Healthy Adult Volunteers To Evaluate The Palatability And Estimate The Bioavailability Of Three Prototype Formulations Of Crizotinib
Brief Title: A Study To Taste Three New Types Of Crizotinib Formulation In Comparison Of An Oral Solution And To Measure The Amount Of Crizotinib In The Body After These Formulations Are Orally Given, Relative To Capsule Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A8081041
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: healthy volunteers; taste; bioavailability
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 will be an open label, randomized, 4 period, 4 treatment, 4 sequence, cross over sensory evaluation of three new prototype formulations (75 mg dose of crizotinib as prototypes 0.529 mg/mg, 0.470 mg/mg and 0.420 mg/mg Microspheres) and OS (75 mg dose of crizotinib)via use of a Crizotinib Taste Assessment - Questionnaire for Cohort 1 in healthy adults.
  Interventions: Drug: Crizotinib prototype microsphere 0.529 mg/mg; Drug: crizotinib prototype microsphere 0.470 mg/mg; Drug: crizotinib prototype microsphere 0.420 mg/mg; Drug: crizotinib oral solution
- Cohort 2 (Experimental): This cohort will be an open label, randomized, 5 period, 5 treatment, 4 sequence, cross over single dose bioavailability study employing administration of four crizotinib formulations Treatments E, F, G and H (Crizotinib 250 mg dose Formulated Capsule and 250 mg dose crizotinib as prototypes 0.529 mg/mg, 0.470 mg/mg and 0.420 mg/mg Microspheres, respectively) in the fasted state to healthy adult subjects (Periods 1-4). In addition, Treatment I (250 mg dose of crizotinib OS) will be administered at Period 5, for a taste evaluation only (no pharmacokinetic (PK) sample collection after the dose), in the period immediately following the completion of Period 4 of Cohort 2. A Crizotinib Taste Assessment - Questionnaire for Cohort 2 will be filled by all subjects.
  Interventions: Drug: crizotinib prototype microsphere 0.529 mg/mg; Drug: crizotinib prototype microsphere 0.470 mg/mg; Drug: crizotinib prototype microsphere 0.420 mg/mg; Drug: crizotinib capsule; Drug: crizotinib oral solution

INTERVENTIONS:
Drug: Crizotinib prototype microsphere 0.529 mg/mg — Subjects will take each sample into their mouths, swirl the sample for approximately 30 seconds, and then expectorate into an empty cup.
  Arms: Cohort 1
Drug: crizotinib prototype microsphere 0.470 mg/mg — Subjects will take each sample into their mouths, swirl the sample for approximately 30 seconds, and then expectorate into an empty cup.
  Arms: Cohort 1
Drug: crizotinib prototype microsphere 0.420 mg/mg — Subjects will take each sample into their mouths, swirl the sample for approximately 30 seconds, and then expectorate into an empty cup.
  Arms: Cohort 1
Drug: crizotinib oral solution — Subjects will take each sample into their mouths, swirl the sample for approximately 30 seconds, and then expectorate into an empty cup.
  Arms: Cohort 1
Drug: crizotinib prototype microsphere 0.529 mg/mg — Subjects will receive a single 250-mg oral dose of crizotinib.
  Arms: Cohort 2
Drug: crizotinib prototype microsphere 0.470 mg/mg — Subjects will receive a single 250-mg oral dose of crizotinib.
  Arms: Cohort 2
Drug: crizotinib prototype microsphere 0.420 mg/mg — Subjects will receive a single 250-mg oral dose of crizotinib.
  Arms: Cohort 2
Drug: crizotinib capsule — Subjects will receive a single 250-mg oral dose of crizotinib.
  Arms: Cohort 2
Drug: crizotinib oral solution — Subjects will receive a single 250-mg oral dose of crizotinib.
  Arms: Cohort 2

SUMMARY:
This study is intended to evaluate the sensory attributes and estimate the relative bioavailability of three prototype oral formulations. Subjects will either taste 75-mg doses by "swirl and spit" (Cohort 1) or will receive five oral single 250-mg doses with a washout period of at least 14 days (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests.
* Female subjects of non child bearing potential must have a Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Pregnant or nursing females; females of childbearing potential.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 3 months
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 3 months
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Maximum Observed Plasma Concentration (Cmax) | 3 months
Overall liking, mouth feel, bitterness, tongue/mouth burn of sensory attributes and formulation preference for Cohort 1 | 3 months

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 3 months
Plasma Decay Half-Life (t1/2) | 3 months
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | 3 months
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 3 months
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed
Overall liking, bitterness, mouth feel, tongue/mouth burn, throat burn of sensory attributes for Cohort 2. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081041&StudyName=A%20Study%20To%20Taste%20Three%20New%20Types%20Of%20Crizotinib%20Formulation%20In%20Comparison%20Of%20An%20Oral%20Solution%20And%20To%20%20Measure%20The%20Amount%20Of%20Crizo